CLINICAL TRIAL: NCT00716963
Title: Does a Lipophilic Steroid Inhaled After an Early Allergic Reaction Affect the Late Reaction?
Brief Title: Does Fluticasone Propionate Reduce the Late Allergic Reaction When the Drug is Given Post-allergen?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: AZ2008lr
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2015-04

CONDITIONS: Mild Intermittent Asthma
Keywords: late allergic response; fluticasone propionate
MeSH Terms: interventions — Fluticasone; Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Fluticasone propionate (Flovent Diskus) 250 mcg
  Interventions: Drug: Fluticasone propionate (Flovent Diskus) 250 mcg
- 2 (Active Comparator): budesonide 400mcg
  Interventions: Drug: budesonide 400 mcg
- 3 (Placebo Comparator): placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fluticasone propionate (Flovent Diskus) 250 mcg — Flovent Diskus 250 mcg
  Other Names: fluticasone propionate Flovent Diskus250 mcg
  Arms: 1
Drug: budesonide 400 mcg — budesonide 400 mcg
  Other Names: Pulmicort Turbuhaler 200 mcg
  Arms: 2
Other: Placebo — Placebo
  Arms: 3

SUMMARY:
The investigators propose a 3-treatment, placebo-controlled, double-dummy, double-blinded, randomized, crossover study in which single doses of placebo, will be compared to Fluticasone propionate (Flovent Diskus) 250 mcg and budesonide 400 mcg administered after allergen challenge, at cessation of the early allergic reaction (at 20% fall in FEV1 from post-allergen peak)

DETAILED DESCRIPTION:
The aim of this pilot study is to evaluate whether fluticasone propionate affects the late allergic reaction after a single dose post-allergen challenge administered following cessation of the early allergic reaction.

Six subjects with mild asthma will be asked to volunteer for the study.The diagnosis of asthma will be and includes the presence of variable airflow limitation and AHR (PC20 methacholine < 16 mg/mL). Subjects will be asked to participate if they demonstrate an allergen-induced early and late asthmatic response of at least 20% and 15% reduction in FEV1, respectively.

The study will consist of 4 periods, composed of a screening allergen period with 3 subsequent allergen challenge/treatment periods. Each period will be separated with a washout of at least 2 weeks. Subjects who demonstrate a dual asthmatic response in the screening period will be selected for randomization to treatment.

ELIGIBILITY:
Inclusion Criteria:

* mild asthma
* nonsmokers
* allergen-induced early and late asthmatic response

Exclusion Criteria:

* no medication other than infrequent ( < twice weekly) inhaled beta2-agonists
* not be exposed to sensitizing allergens
* asthma exacerbation or respiratory tract infection in the past4 weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2008-07; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul O'Byrne, MD, Principal Investigator — McMaster University; Gail Gauvreau, PhD, Study Director — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Bousquet J, Clark TJ, Hurd S, Khaltaev N, Lenfant C, O'byrne P, Sheffer A. GINA guidelines on asthma and beyond. Allergy. 2007 Feb;62(2):102-12. doi: 10.1111/j.1398-9995.2006.01305.x. PMID 17298416
- [Background] Gauvreau GM, Doctor J, Watson RM, Jordana M, O'Byrne PM. Effects of inhaled budesonide on allergen-induced airway responses and airway inflammation. Am J Respir Crit Care Med. 1996 Nov;154(5):1267-71. doi: 10.1164/ajrccm.154.5.8912734.
- [Background] Paggiaro PL, Dente FL, Morelli MC, Bancalari L, Di Franco A, Giannini D, Vagaggini B, Bacci E, Fabbri LM, Giuntini C. Postallergen inhaled budesonide reduces late asthmatic response and inhibits the associated increase of airway responsiveness to methacholine in asthmatics. Am J Respir Crit Care Med. 1994 Jun;149(6):1447-51. doi: 10.1164/ajrccm.149.6.8004297.
- [Background] Duong M, Gauvreau G, Watson R, Obminski G, Strinich T, Evans M, Howie K, Killian K, O'Byrne PM. The effects of inhaled budesonide and formoterol in combination and alone when given directly after allergen challenge. J Allergy Clin Immunol. 2007 Feb;119(2):322-7. doi: 10.1016/j.jaci.2006.10.018. Epub 2006 Dec 4. PMID 17141859
- [Background] Cockcroft DW, McParland CP, O'Byrne PM, Manning P, Friend JL, Rutherford BC, Swystun VA. Beclomethasone given after the early asthmatic response inhibits the late response and the increased methacholine responsiveness and cromolyn does not. J Allergy Clin Immunol. 1993 Jun;91(6):1163-8. doi: 10.1016/0091-6749(93)90319-b. PMID 8509579
- [Background] Boulet LP, Gauvreau G, Boulay ME, O'Byrne P, Cockcroft DW; Clinical Investigative Collaboration, Canadian Network of Centers of Excellence AllerGen. The allergen bronchoprovocation model: an important tool for the investigation of new asthma anti-inflammatory therapies. Allergy. 2007 Oct;62(10):1101-10. doi: 10.1111/j.1398-9995.2007.01499.x. PMID 17845579
- [Background] Gauvreau GM, Boulet LP, Hessel EM, Watson RM, Milot J, Coffman RL, et al. A phase 2, randomized, observer-blind, placebo-controlled study of the efficacy, safety and tolerability of inhaled 1018 ISS immunostimulatory oligonucleotide in subjects with mild to moderate asthma. Am.J.Respir.Crit Care Med. 171, A81. 2005. Ref Type: Abstract
- [Background] Cockcroft DW, Murdock KY, Kirby J, Hargreave F. Prediction of airway responsiveness to allergen from skin sensitivity to allergen and airway responsiveness to histamine. Am Rev Respir Dis. 1987 Jan;135(1):264-7. doi: 10.1164/arrd.1987.135.1.264. PMID 3800152
- [Background] Cockcroft DW, Davis BE, Boulet LP, Deschesnes F, Gauvreau GM, O'Byrne PM, Watson RM. The links between allergen skin test sensitivity, airway responsiveness and airway response to allergen. Allergy. 2005 Jan;60(1):56-9. doi: 10.1111/j.1398-9995.2004.00612.x. PMID 15575931
- [Background] Pizzichini E, Pizzichini MM, Efthimiadis A, Evans S, Morris MM, Squillace D, Gleich GJ, Dolovich J, Hargreave FE. Indices of airway inflammation in induced sputum: reproducibility and validity of cell and fluid-phase measurements. Am J Respir Crit Care Med. 1996 Aug;154(2 Pt 1):308-17. doi: 10.1164/ajrccm.154.2.8756799.
- [Background] O'Byrne PM, Dolovich J, Hargreave FE. Late asthmatic responses. Am Rev Respir Dis. 1987 Sep;136(3):740-51. doi: 10.1164/ajrccm/136.3.740. No abstract available. PMID 3115156
- [Background] Inman MD, Watson R, Cockcroft DW, Wong BJ, Hargreave FE, O'Byrne PM. Reproducibility of allergen-induced early and late asthmatic responses. J Allergy Clin Immunol. 1995 Jun;95(6):1191-5. doi: 10.1016/s0091-6749(95)70075-7. PMID 7797787
- [Background] Gauvreau GM, Watson RM, Rerecich TJ, Baswick E, Inman MD, O'Byrne PM. Repeatability of allergen-induced airway inflammation. J Allergy Clin Immunol. 1999 Jul;104(1):66-71. doi: 10.1016/s0091-6749(99)70115-6. PMID 10400841

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluticasone/Budesonide/Placebo: Subjects receive Fluticasone after early allergic response induced by allergen challenge. At least 2 week wash out period. Subjects receive Budesonide after early allergic response induced by allergen challenge. At least 2 week wash out period. Subjects receive placebo after early allergic response induced by allergen challenge.
- Fluticasone/Placebo/Budesonide: Subjects receive Fluticasone after early allergic response induced by allergen challenge. At least 2 week wash out period. Subjects receive placebo after early allergic response induced by allergen challenge. At least 2 week wash out period. Subjects receive Budesonide after early allergic response induced by allergen challenge.
- Budesonide/Fluticasone/Placebo: Subjects receive Budesonide after early allergic response induced by allergen challenge. At least 2 week wash out period. Subjects receive Fluticasone after early allergic response induced by allergen challenge. At least 2 week wash out period. Subjects receive placebo after early allergic response induced by allergen challenge.
- Budesonide/Placebo/Fluticasone: Subjects receive Budesonide after early allergic response induced by allergen challenge. At least 2 week wash out period. Subjects receive placebo after early allergic response induced by allergen challenge. At least 2 week wash out period. Subjects receive Fluticasone after early allergic response induced by allergen challenge.
- Placebo/Fluticasone/Budesonide: Subjects receive placebo after early allergic response induced by allergen challenge. At least 2 week wash out period. Subjects receive Fluticasone after early allergic response induced by allergen challenge. At least 2 week wash out period. Subjects receive Budesonide after early allergic response induced by allergen challenge.
- Placebo/Budesonide/Fluticasone: Subjects receive placebo after early allergic response induced by allergen challenge. At least 2 week wash out period. Subjects receive Budesonide after early allergic response induced by allergen challenge. At least 2 week wash out period. Subjects receive Fluticasone after early allergic response induced by allergen challenge.
Period: Overall Study
Arm/Group | Fluticasone/Budesonide/Placebo | Fluticasone/Placebo/Budesonide | Budesonide/Fluticasone/Placebo | Budesonide/Placebo/Fluticasone | Placebo/Fluticasone/Budesonide | Placebo/Budesonide/Fluticasone
Started | 2 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Screening/Baseline Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: The Magnitude of the Early Asthmatic Response, Expressed as a Percentage Change in FEV1.
Time Frame: Before inhalation 3 hours
Population: Instead of re-listing participant flow, data was taken from each subject arm and re-listed here as the 3 arms each subject underwent.
Measure: Mean (Standard Deviation); unit: percentage fall FEV1
Arm/Group | Fluticasone Propionate (Flovent Diskus) 250 mcg | Budesonide 400mcg | Placebo
Number analyzed (Participants) | 6 | 6 | 6
percentage fall FEV1 | -30.5 (9.3) | -39.0 (12.3) | -31.9 (10.6)

2. Primary Outcome: The Magnitude of the Late Asthmatic Response, Expressed as a Percentage Change in FEV1.
Time Frame: 7 hours after challenge
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage fall FEV1
Arm/Group | Fluticasone Propionate (Flovent Diskus) 250 mcg | Budesonide 400mcg | Placebo
Number analyzed (Participants) | 6 | 6 | 6
percentage fall FEV1 | -11.6 (14.2) | -14.7 (6.6) | -24 (7.2)

3. Secondary Outcome: The Magnitude of Allergen-induced Airway Hyperresponsiveness (Methacholine PC20) and Inflammation (Sputum Eosinophils).
Time Frame: Before inhalation both evaluations (0 hours)
Reporting Status: Not Posted

4. Secondary Outcome: The Magnitude of Allergen-induced Airway Hyperresponsiveness (Methacholine PC20) and Inflammation (Sputum Eosinophils)
Time Frame: sputum @ 7 hours
Reporting Status: Not Posted

5. Secondary Outcome: The Magnitude of Allergen-induced Airway Hyperresponsiveness (Methacholine PC20) and Inflammation (Sputum Eosinophils)
Time Frame: 24 hours methacholine and sputum
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Fluticasone Propionate (Flovent Diskus) 250 mcg | Budesonide 400mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days